CLINICAL TRIAL: NCT00005188
Title: Quantitative Genetic Analysis of Lipid Research Clinic Family Data
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 1066; R01HL033973 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2004-08

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Coronary Disease; Tangier Disease; Atherosclerosis
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Coronary Disease; Tangier Disease; Atherosclerosis

SUMMARY:
To assess the mode of inheritance of familial combined hyperlipidemia and familial primary hypoalphalipoproteinemia and to resolve genetic and familial environmental effects on several phenotypes of importance to coronary heart disease.

DETAILED DESCRIPTION:
BACKGROUND:

Although coronary heart disease has long been known to aggregate in families, in 1986 little was known about the relative importance of genetic and environmental factors. This was partly due to the heterogeneous nature of the disease. Instead of analyzing complex endpoints, the tendency had been to focus on the individual risk factors or phenotypes. Plasma lipids and lipoproteins are heterogeneous risk factors that have been analyzed as subgroups from a genetic epidemiological perspective. Attention turned to the familial aggregation of risk factors, particularly the hyperlipidemias, hypertension, and diabetes.

In 1971, the National Heart and Lung Institute began a series of epidemiologic studies at several North American sites under the Lipid Research Clinics Program. The Family Study was designed to investigate the familial association of blood lipids, lipoproteins, and dyslipoproteinemias. This study complemented and did not duplicate ongoing analysis of Lipid Research Clinics data.

DESIGN NARRATIVE:

The study addressed seven phenotypes, all derived from fasting blood samples: total cholesterol, total triglyceride, LDL-cholesterol, HDL-cholesterol, VLDL-cholesterol, uric acid, and glucose levels. The data had already been collected at Lipid Research Clinics in Cincinnati, Iowa, Oklahoma, Minneapolis, and Stanford. Univariate and bivariate segregation analysis were conducted on the mode of inheritance of familial combined hyperlipidemia and familial primary hypoalphalipoproteinemia. Path analysis was used to resolve cultural and biological inheritance for each phenotype within each clinic and for resolution of population heterogeneity among the five Lipid Research Clinics. A general bivariate path model was used to analyze the associations among the various phenotypes. General models were used to analyze temporal trends in family resemblance for the seven phenotypes.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1986-07; Study Completion 1991-06 (Actual)

REFERENCES:
- [Background] Rao DC, Wette R. Nonrandom sampling in genetic epidemiology: maximum likelihood methods for multifactorial analysis of quantitative data ascertained through truncation. Genet Epidemiol. 1987;4(5):357-76. doi: 10.1002/gepi.1370040505. PMID 3319764
- [Background] Rao DC, Vogler GP, McGue M, Russell JM. Maximum-likelihood estimation of familial correlations from multivariate quantitative data on pedigrees: a general method and examples. Am J Hum Genet. 1987 Dec;41(6):1104-16. PMID 3687943
- [Background] Rao DC, Wette R, Ewens WJ. Multifactorial analysis of family data ascertained through truncation: a comparative evaluation of two methods of statistical inference. Am J Hum Genet. 1988 Mar;42(3):506-15. PMID 3348215
- [Background] Wette R, McGue MK, Rao DC, Cloninger CR. On the properties of maximum likelihood estimators of familial correlations under variable sibship size. Biometrics. 1988 Sep;44(3):717-25. PMID 3203127
- [Background] Province MA, Rao DC. Familial aggregation in the presence of temporal trends. Stat Med. 1988 Jan-Feb;7(1-2):185-98. doi: 10.1002/sim.4780070120. PMID 3258435
- [Background] Borecki IB, Laskarzewski P, Rao DC. Genetic factors influencing apolipoprotein AI and AII levels in a kindred with premature coronary heart disease. Genet Epidemiol. 1988;5(6):393-406. doi: 10.1002/gepi.1370050604. PMID 3145239
- [Background] Province MA, Tishler P, Rao DC. Repeated-measures model for the investigation of temporal trends using longitudinal family studies: application to systolic blood pressure. Genet Epidemiol. 1989;6(2):333-47. doi: 10.1002/gepi.1370060204. PMID 2721928
- [Background] McGue M, Wette R, Rao DC. Path analysis under generalized marital resemblance: evaluation of the assumptions underlying the mixed homogamy model by the Monte Carlo method. Genet Epidemiol. 1989;6(2):373-88. doi: 10.1002/gepi.1370060207. PMID 2721930
- [Background] Reddy BM, Rao DC. Phenylthiocarbamide taste sensitivity revisited: complete sorting test supports residual family resemblance. Genet Epidemiol. 1989;6(3):413-21. doi: 10.1002/gepi.1370060304. PMID 2753351
- [Background] Rao DC, Wette R. Nonrandom sampling in genetic epidemiology: an implementation of the Hanis-Chakraborty method for multifactorial analysis. Genet Epidemiol. 1989;6(3):461-70. doi: 10.1002/gepi.1370060308. PMID 2753354
- [Background] Perusse L, Rice T, Bouchard C, Vogler GP, Rao DC. Cardiovascular risk factors in a French-Canadian population: resolution of genetic and familial environmental effects on blood pressure by using extensive information on environmental correlates. Am J Hum Genet. 1989 Aug;45(2):240-51. PMID 2757030
- [Background] Byard PJ, Mukherjee BN, Bhattacharya SK, Russell JM, Rao DC. Familial aggregation of blood pressure and anthropometric variables in patrilocal households. Am J Phys Anthropol. 1989 Jul;79(3):305-11. doi: 10.1002/ajpa.1330790306. PMID 2764083
- [Background] McGue M, Gerrard JW, Lebowitz MD, Rao DC. Commingling in the distributions of immunoglobulin levels. Hum Hered. 1989;39(4):196-201. doi: 10.1159/000153860. PMID 2583731
- [Background] Rao DC, Wette R. Environmental index in genetic epidemiology: an investigation of its role, adequacy, and limitations. Am J Hum Genet. 1990 Jan;46(1):168-78. PMID 2294748
- [Background] Vogler GP, Wette R, Laskarzewski PM, Perry TS, Rice T, Province MA, Rao DC. Heterogeneity in the biological and cultural determinants of high-density lipoprotein cholesterol in five North American populations: the Lipid Research Clinics Family Study. Hum Hered. 1989;39(5):249-57. doi: 10.1159/000153868. PMID 2613250
- [Background] Rice T, Vogler GP, Perry TS, Laskarzewski PM, Province MA, Rao DC. Heterogeneity in the familial aggregation of fasting serum uric acid level in five North American populations: the Lipid Research Clinics Family Study. Am J Med Genet. 1990 Jun;36(2):219-25. doi: 10.1002/ajmg.1320360216. PMID 2368810
- [Background] Rice T, Vogler GP, Perry TS, Laskarzewski PM, Province MA, Rao DC. Heterogeneity in the familial aggregation of fasting plasma glucose in five North American populations: the Lipid Research Clinics Family Study. Int J Epidemiol. 1990 Jun;19(2):290-6. doi: 10.1093/ije/19.2.290. PMID 2198234
- [Background] Rice T, Laskarzewski PM, Rao DC. Commingling and complex segregation analysis of fasting plasma glucose in the Lipid Research Clinics family study. Am J Med Genet. 1992 Nov 1;44(4):399-404. doi: 10.1002/ajmg.1320440402. PMID 1442875
- [Background] Rice T, Laskarzewski PM, Perry TS, Rao DC. Commingling and segregation analysis of serum uric acid in five North American populations: the Lipid Research Clinics family study. Hum Genet. 1992 Sep-Oct;90(1-2):133-8. doi: 10.1007/BF00210757. PMID 1427769
- [Background] Rice T, Vogler GP, Laskarzewski PM, Perry TS, Rao DC. Familial aggregation of lipids and lipoproteins in families ascertained through random and nonrandom probands in the Minnesota Lipid Research Clinic Family Study. Hum Biol. 1991 Aug;63(4):419-39. PMID 1889794
- [Background] Rice T, Vogler GP, Laskarzewski PM, Perry TS, Rao DC. Familial aggregation of lipids and lipoproteins in families ascertained through random and nonrandom probands in the Stanford Lipid Research Clinics Family Study. Am J Med Genet. 1991 Jun 1;39(3):270-7. doi: 10.1002/ajmg.1320390306. PMID 1867276
- [Background] Rice T, Vogler GP, Perry TS, Laskarzewski PM, Rao DC. Familial aggregation of lipids and lipoproteins in families ascertained through random and nonrandom probands in the Iowa Lipid Research Clinics family study. Hum Hered. 1991;41(2):107-21. doi: 10.1159/000153987. PMID 1855782
- [Background] Borecki IB, Rao DC, Yaouanq J, Lalouel JM. Serum ferritin as a marker of affection for genetic hemochromatosis. Hum Hered. 1990;40(3):159-66. doi: 10.1159/000153924. PMID 2365376
- [Background] Vogler GP, Wette R, McGue MK, Rao DC. Properties of alternative estimators of familial correlations under variable sibship size. Biometrics. 1995 Mar;51(1):276-83. PMID 7766782